CLINICAL TRIAL: NCT00245453
Title: Randomized Aseptic Pharmacokinetic Pharmacodynamic Outpatient Registry Trial of Respiratory Tract Infections in Adults (RAPPORT)
Brief Title: Outpatient Registry Trial of Respiratory Tract Infections in Adults
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: CPL Associates (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A6004
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Pneumonia, Bacterial; Bronchitis, Chronic
Keywords: pneumonia; Spneumoniae; bronchitis; telithromycin; azithromycin
MeSH Terms: conditions — Pneumonia, Bacterial; Bronchitis, Chronic; Pneumonia; Bronchitis | interventions — Azithromycin; telithromycin

ARMS (3):
- 1 Azithromycin (Active Comparator)
  Interventions: Drug: azithromycin
- 2 Clarythromycin (Active Comparator)
  Interventions: Drug: Clarythromycin
- 3 Telithromycin (Active Comparator)
  Interventions: Drug: telithromycin

INTERVENTIONS:
Drug: azithromycin — 250 mg tablets; 2 tablets on day 1 (500 mg load) and 1 tablet QD on days 2-5
  Arms: 1 Azithromycin
Drug: telithromycin — 400 mg tablets; 2 tablets once daily (QD) for 5 days
  Arms: 3 Telithromycin
Drug: Clarythromycin — 500 mg extended release tablets; 2 tablets QD for 7 days
  Arms: 2 Clarythromycin

SUMMARY:
To measure the speed of bacterial eradication from the respiratory tract after administration of azithromycin or telithromycin.

DETAILED DESCRIPTION:
To Evaluate the relationship between rate of S. pneumoniae killing in sputum, PK/PD, and clinical response of oral telithromycin and azithromycin in patients with AECB or CAP and to determine if there is a difference in the rates of infection site bacterial killing (as described above) between these 3 antibiotics against penicillin- and erythromycin-resistant S.pneumoniae

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, either males or non-pregnant females, aged 18 to 75 years of age with clinical findings of CAP or AECB who are amenable to serial nasopharyngeal and oropharyngeal sampling and having positive Binax-NOW tests indicating infection with Streptococcus pneumoniae
* Patients with a medical history and clinical findings consistent with a respiratory tract infection. A patient with advanced COPD, repeated exacerbations by history, a BINAX-NOW test consistent with S. pneumoniae and/or proven culture positivity for S. pneumoniae may be enrolled
* All patients (CAP or AECB) must produce purulent sputum and be positive on the Urinary BINAX-NOW assay.
* The female patient of child bearing potential must agree to use an accepted method of contraception (i.e., oral or implanted contraceptive with a barrier method, spermicide and barrier methods, or IUD). The patient must agree to continue with the same method throughout the study.

Exclusion Criteria:

* Baseline sputum cultures known to be negative for S. pneumoniae, or negative urinary BINAX-NOW.
* Patients with a microbiologically documented pathogen known prior to inclusion to be resistant to any of the study medications.
* History of hypersensitivity to macrolides, azalides, ketolide antibiotics or history of serious hypersensitivity reaction to any drug.
* Pre-existing impaired hepatic function or impaired renal function CCL <20ml/min
* Patients who will require on-study treatment with medications known to have contraindicated drug interactions with telithromycin
* Treatment with more than one dose of an antimicrobial prior to entry into the study

Others as per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Time to bacterial eradication | 11-18 days
Bacteriologic outcome | 11-18 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerome J Schentag, Pharm.D., Principal Investigator — State University of New York at Buffalo; Joseph Paladino, Pharm.D., Study Director — State University of New York at Buffalo
Locations (2):
- United States (2):
  - Western Kentucky Pulmonary Clinic, Louisville, Kentucky
  - Northshore Research Associates, Slidell, Louisiana

REFERENCES:
- See also: Related Info — http://www.cplassociates.com